CLINICAL TRIAL: NCT04804696
Title: Toripalimab with Paclitaxel and Cisplatin As Neoadjuvant Treatment for Esophageal Squamous Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Several clinical trials had showed that anti-PD-1 agents combined with chemotherapy as neoadjuvant treatment could increase pCR rate in 2024. In order to protect the interest of patients, this trial was stopted.
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Xiaodong Zhang, Dean of VIP2 Gastrointestinal Cancer Division of Medical Department, Beijing Cancer Hospital, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESCC003
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Esophageal Squamous Cell Cancer
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — toripalimab; Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TPC treatment (Experimental): Neoadjuvant treatment of toripalimab, paclitaxel and cisplatin
  Interventions: Drug: Toripalimab; Drug: Paclitaxel; Drug: Cisplatin

INTERVENTIONS:
Drug: Toripalimab — Patients received toripalimab 240 mg I.V. drip on days 1 and 22.
  Other Names: JS001; TAB001
Drug: Paclitaxel — Patients received paclitaxel of 175mg/m2 I.V. drip on days 1 and 22.
Drug: Cisplatin — Patients received cisplatin of 70mg/m2 I.V. drip on days 1 and 22.

SUMMARY:
Neoadjuvant chemoradiotherapy or chemotherapy followed by surgery is the standard treatment for local advanced esophageal cancer (EC). It had been demonstrated that patients who achieve pathologic complete response (pCR) after neoadjuvant treatment had better prognosis. However, the pCR rate were about only 5-10% in neoadjuvant chemotherapy and 20-40% in neoadjuvant concurrent chemoradiotherapy.

PD-1 antibody based immunotherapy alone as second-line treatment or combined with chemotherapy as first-line treatment had been proved that could prolong overall survival of EC patients. And a recent phase 3 clinical trial CheckMate 577 reported that, as adjuvant treatment, nivolumab could improve disease-free survival in EC and esophageal-gastric junction cancer.

The aim of this study was to evaluate the efficacy and safety of toripalimab, an anti-PD-1 antibody, combined with paclitaxel and cisplatin as neoadjuvant treatment in local advanced esophageal squamous cell carcinoma (ESCC). We hope this combining treatment would increase the pCR rate of neoadjuvant chemotherapy and improve survival of patients, and at the menatime avoid the adverse events of neoadjuvant radiotherapy. This study will provide valuable information for further clinical trials of both Toripalimab and other immune checkpoint inhibition agents in treatment of esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70 years old, both gender.
2. Histopathologically confirmed esophageal squamous cell carcinoma.
3. No previous chemotherapy, radiotherapy, traditional Chinese medicine and other anti-tumor treatments.
4. Imaging (CT or MR) or ultrasound endoscopy confirmed local advanced resectable lesions ( AJCC 8th edition standard, stage 3N0M0 or T1-4aN+M0).
5. The ECOG performance status score of 0-1.
6. Normal functionof all major organs, that is:

   * Hemoglobin (Hb) ≥ 100g/L,

     * Neutrophils (ANC) ≥ 1.5×109/L, ③ Platelet count (PLT) ≥100×109/L, ④ Prothrombin time (PT) and partial prothrombin time (PTT) ≤ 1.5×upper limit of normal (ULN). (For the use of a stable dose of anticoagulant therapy such as low molecular weight heparin or warfarin, if the INR is within the expected therapeutic range of anticoagulants, patient could be screened); ⑤ Serum creatinine (Cr) ≤ 1.5 ×ULN, or 24-hour creatinine clearance rate >60mL/min（Cockcroft-Gault）; ⑥ Total blood bilirubin (TB) ≤ 1.5ULN; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5×ULN; albumin (ALB) ≥ 30g/L.
7. The cardiac function is basically normal, the left ventricular ejection fraction is ≥50%, and the blood pressure is under controlled within 140/90 mmHg before enrollment.
8. Pulmonary function is basically normal, without moderate to severe obstructive and diffuse dysfunction.
9. Be able to provide tissue samples for biomarkers analysis, such as PD-L1 expression.
10. Women of childbearing age must have taken reliable contraceptive measures or undergo a pregnancy test (serum) within 7 days before enrollment, and the result is negative, and are willing to use appropriate methods of contraception. For men, they must agree to use appropriate methods of contraception or have been surgically sterilized during the trial period and within 8 weeks after the last trial drug administration;
11. Voluntarily sign an informed consent form (or signed by a legal representative) to prove that they understand the purpose of the research and the operations required by the research and are willing to participate in the research.

Exclusion Criteria:

1. Adenocarcinoma, small cell carcinoma, and other non-squamous cell carcinoma types of esophageal cancer.
2. Imaging examinations (CT or MRI) or endoscopic ultrasonography revealed early stage esophageal cancer, including: carcinoma in situ (Tis), lesions only invaded the mucosa layer or the muscularis propria without lymph node metastasis (T1-2N0).
3. Imaging examinations (CT or MRI) revealed unresectable disease including invasion of vertebral body, aorta, and organs (T4b), or with distant metastases such as lungs, liver, bones and other organ metastases (M1) ;
4. Imaging (esophagography, CT or MR) examination within 4 weeks before enrollment revealed esophageal mediastinal fistula or esophagotracheal fistula.
5. Gastrointestinal bleeding such as hematemesis or melena within 4 weeks before the first dose of treatment.
6. Allergic to PD-1 antibodies, paclitaxel, or cisplatin.
7. Receiving previous anti-tumor treatments such as chemotherapy, radiotherapy, molecular targeted therapy, or Chinese medicine treatment within 4 weeks before enrollment.
8. Receiving corticosteroids (>10 mg prednisone or equivalent dose per day) or other immunosuppressive therapy within 2 weeks before enrollment, except for those who use corticosteroids to prevent allergies, nausea, and vomiting.
9. Received live vaccines within 4 weeks before the first dose of treatment.
10. Receiving major surgery or suffered severe trauma within 4 weeks before the first dose of treatment.
11. Complicated with active autoimmune diseases, or history of autoimmune diseases (such as interstitial pneumonia, colitis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, hypothyroidism, including but Not limited to these diseases or syndromes). Except: vitiligo, cured childhood asthma/allergic adults without any intervention, autoimmune-mediated hypothyroidism treated with a stable dose of thyroid replacement hormone, and type I diabetes with a stable dose of insulin.
12. A history of immunodeficiency, including HIV positive, acquired or congenital immunodeficiency diseases, organ transplantation, or bone marrow transplantation.
13. With clinical symptoms of cardiovascular diseases which were not well controlled, including but not limited to: heart failure above NYHA II; unstable angina; myocardial infarction within 1 year; clinically significant supraventricular or ventricular arrhythmia and is still uncontrolled without clinical intervention or clinical intervention;
14. Severe infections (CTC AE> Grade 2) occurred within 4 weeks before the first dose of treatment, such as severe pneumonia, bacteremia, infectious comorbidities that require hospitalization, etc.; baseline chest imaging examinations suggest the presence of active lungs Inflammation; having symptoms and signs of infection or taken oral or intravenous antibiotic treatment within 2 weeks before the first dose of treatment except for prophylactic use of antibiotics.
15. A history of interstitial lung disease and a history of non-infectious pneumonia.
16. With active pulmonary tuberculosis infection identified by medical history or CT examination, or a history of active pulmonary tuberculosis infection within 1 year before enrollment.
17. Active hepatitis B (quantity of HBV DNA ≥100 IU/mL), or hepatitis C (hepatitis C antibody is positive, and HCV-RNA is higher than the lower limit of the analytical method) infection.
18. Complicated with chronic nephritis, or urine routine test indicates urine protein ≥ ++, or 24-hour urine protein ≥ 1.0 g.
19. Abnormal blood coagulation function (INR or PT or PTT> 1.5 ULN), potential risk of bleeding, or receiving thrombolysis or anticoagulation therapy;
20. With other malignant tumor diagnosed within 5 years before the first dose of treatment. Exclude malignant tumors with low risk of metastasis and death, such as fully treated basal cell or squamous cell skin cancer or cervical carcinoma in situ.
21. Women who are pregnant or breastfeeding.
22. According to the researcher's judgment, there are other factors that may lead to forced termination. Such as suffering from other serious diseases (including mental illness) requiring combined treatment, significant abnormal laboratory test values, or family or social factors, etc., may affect the safety of subjects or the collection of experimental data.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
Pathologic complete response rate | Three weeks after surgery of last enrolled subject. Estimate up to 2 years
  The rate of pathologic complete response rate after neoadjuvant therapy.

SECONDARY OUTCOMES:
Objective Response Rate | One month after 2 cycles' treatment of last enrolled subject. Estimate up to 2 years
  The percentage of patients having a complete response or a partial response to protocol treatment. Objective response will be measured by RECIST 1.1.
R0 resection rate | Three weeks after surgery of last enrolled subject. Estimate up to 2 years
  The R0 resection rate of esophagectomy
Major pathologic response rate | Three weeks after surgery of last enrolled subject. Estimate up to 2 years.
  The percentage of subjects with ≤10% survival tumor cells in the resected specimens after neoadjuvant therapy accounted for all subjects who received surgical treatment.
Disease-free survival | From date of surgery until the date of death from any cause or the date of first documented disease progression whichever came first. Estimate up to three years.
  The time from enrollment to recurrence of tumor or death.
Overall survival | From enrollment to death of patients. Estimate up to 5 years.
  The length of time from enrollment until the time of death
Adverse events | From enrollment to 60 days after the end protocol treatment
  The incidence of adverse events and the incidence of severe adverse events（ grade 3-4) .

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital / Peking University Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No